CLINICAL TRIAL: NCT03416452
Title: Gait Disorders in Parkinson's Disease
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator left the NIH.
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 180050; 18-N-0050
Record Dates: First submitted 2018-01-30; First posted 2018-01-31 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Parkinson's Disease
Keywords: Gait; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- PD patients no (Experimental): PD patients without freezing of gait
  Interventions: Device: Mobile Gait Trainer
- Healthy (Placebo Comparator): HV using Mobile Gait Trainer
  Interventions: Device: Mobile Gait Trainer
- PD patients (Experimental): pd patients using vibratory cueing device
  Interventions: Device: vibratory cueing device
- PD patients 1 (Experimental): PD patients with freezing of gait
  Interventions: Device: vibratory cueing device
- Healthy Volunteers (Experimental): Age and gender matched healthy volunteers.
  Interventions: Device: Mobile Gait Trainer

INTERVENTIONS:
Device: vibratory cueing device — ankle brace with vibrator that provides electric stimulus
  Arms: PD patients; PD patients 1
Device: Mobile Gait Trainer — standard rolling walker that has a battery operated sensor attached to the side, designed to detect footsteps
  Arms: Healthy; Healthy Volunteers; PD patients no

SUMMARY:
Background:

Parkinson s disease (PD) is a neurologic disorder that causes slowness, tremor, rigidity, and imbalance. Gait impairment is also common. There are 2 substudies: (1) Physiology of Freezing and Gait; (2) Vibratory Cueing. Healthy participants can join only Substudy 1.

Objective:

To study gait disorders in PD. Also, to test the effect of specific interventions for gait in people with PD.

Eligibility:

People ages 18 and older who:

Have PD with bilateral symptoms but can walk without a cane or walker

Are healthy

Design:

Participants will be screened in Protocols 93-N-0202 and 01-N-0206.

Both substudies include a physical exam and medical history.

Substudy 1:

Participants will have one 6-hour visit. They must wear a tank tops and shorts with tennis shoes during the visit. They will perform gait tasks. Markers placed on the skin will record movements. They will have an EEG: They will wear an electrode cap to record brain waves. They will wear special glasses to record eye movements. Participants with PD will hold their morning dose of PD drugs. They can choose to be admitted to the hospital the previous evening. Otherwise someone else or a taxi must bring them to the visit. They will first perform the study tasks off their drugs. Then they will take their drugs and repeat them.

Substudy 2:

Participants will have one 3-hour visit. A small vibratory device will be attached to their ankle. Reflective markers placed on the skin will record movements while they walk:

Without the device

With the device, but the vibrator off

With the device, with the vibrator on

With a magnet attached to the ankle

DETAILED DESCRIPTION:
The objective of this protocol is to study the physiology of gait disorders in Parkinson s disease as well as to test the effect of non-invasive interventions on gait function in patients with Parkinson s disease. To this end, this protocol will consist of two sub studies:

1. Sub Study 1: Physiology of Freezing of Gait in Parkinson Disease (abbrev: Physiology of FOG)

   1. Objective: To explore temporospatial gait parameters and joint kinematic patterns in patients with Parkinson disease and freezing of gait. In addition, tracking of eye movements and EEG patterns will also be studied in patients with Parkinson disease and freezing of gait.
   2. Study Population: 15 PD patients with freezing of gait, 15 patients without freezing of gait, 15 age and gender matched healthy volunteers
   3. Design: Prospective Exploratory study
   4. Outcome Measures: Phase variability and coherence of oscillating axial and appendicular components of gait in patients with PD and freezing of gait, visual gaze fixations and saccades during freezing or freezing-like events and when approaching a variable width doorway, EEG patterns during an episode of freezing of gait or freeze-like event. The study will also aim to look at the difference in the phenomenon of FOG in OFF and ON states.
2. Sub Study 2: Effects of Rhythmic Vibratory Cueing to Improve Step Parameters in Parkinson Disease (abbrev. Vibratory Cueing)

   1. Objective: To study changes in gait variables of patients with PD by providing rhythmic vibratory stimuli at the ankle on one limb at preset parameters.
   2. Study population: 15 patients diagnosed as having Parkinson s Disease, Hoehn and Yahr stage 2-3.
   3. Design: Prospective interventional hypothesis testing study. We will evaluate the effects of rhythmic vibratory cueing on gait variables in PD. The effects of vibratory cueing will be tested compared to baseline gait variables and with the use of a magnet (which will be the open label placebo intervention to account to some extent, for the open label design).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years or older
* Able to provide informed consent
* Clinical diagnosis of Parkinson disease by U.K. Parkinson Society Brain Bank Criteria
* Patients must be stage II -III on the Hoehn and Yahr scale

EXCLUSION CRITERIA:

* MoCA<25 within the last 6 months
* Uncontrolled medical condition requiring immediate treatment that would make a walking trial unsafe for the subject.
* Peripheral neuropathy that severely limits gait
* Current or recent orthopedic disorder that severely limits gait
* Current uncontrolled depression or major depressive episode
* Gait disorders other than PD.
* Cannot walk safely without corrective lenses and without support.
* Unable to abstain from PD medications overnight for at least 12 hours before testing
* History of deep brain stimulation surgery
* Subjects who are NINDS employees
* In addition to the preceding criteria, healthy volunteers must also have a normal neurological examination performed within the last year. Healthy volunteers will be healthy subjects without any major medical and neurological or psychiatric disorders established by history and physical/neurological examination. They will also have no gait disorders from any medical or surgical problems as per clinical assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
To examine the relative phase variability or coherence between oscillating axial and appendicular components of gait in PD + FOG, compared to PD-FOG and healthy controls. | ongoing
Changes in Stride length | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Hussain I Merchant, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)

REFERENCES:
- [Background] Kelly VE, Eusterbrock AJ, Shumway-Cook A. The effects of instructions on dual-task walking and cognitive task performance in people with Parkinson's disease. Parkinsons Dis. 2012;2012:671261. doi: 10.1155/2012/671261. Epub 2012 Dec 29. PMID 23326758